CLINICAL TRIAL: NCT00748696
Title: Combined Effects of Resistance Training and Nutritional Supplements in the Treatment of Sarcopenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 06-API-04
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2009-06

CONDITIONS: Sarcopenia
Keywords: sarcopenia; elderly; resistance training; oral nutritional supplement
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention): No intervention
- 2 (Experimental): patient receiving oral nutrition supplement
  Interventions: Dietary Supplement: Fortimel Extra®
- 3 (Experimental): resistance training
  Interventions: Other: resistance training
- 4 (Experimental): patients receiving resistance training and oral nutritional supplement
  Interventions: Other: combined treatment

INTERVENTIONS:
Dietary Supplement: Fortimel Extra® — 260kcal and 20g protein per day
  Arms: 2
Other: resistance training — 3 sessions of resistance training per week
  Arms: 3
Other: combined treatment — 260kcal and 20g protein per day 3 sessions of resistance training per week
  Arms: 4

SUMMARY:
Age-related sarcopenia is associated with increased morbidity, mortality, disability and reduced resistance to metabolic stress. The aim of this study is to assess the effects of resistance training, associated or not with oral nutritional supplements, on skeletal muscle mass in sarcopenic subjects. This is a prospective randomised controlled single-centre study that will last two years, three months for a participant.

200 healthy elderly (70-80 years old) subjects will be screened for sarcopenia by dual energy X-ray absorptiometry. 128 sarcopenic subjects will be randomized into 4 groups:

* group 1: controls
* group 2: oral nutritional supplement (260 kcal and 20 g protein per day)
* group 3: resistance training (3 times per week)
* group 4: oral nutritional supplement + resistance training

Every subject will be assessed at the beginning and at the end of 12 weeks of intervention on:

* muscle mass (DXA)
* muscle function (dynamometers)
* hormonal (testosterone, GH, IGF-1, cortisol) and inflammatory (IL-6, TNF-alpha) profiles
* food intake. Ten subjects in group 4 will undergo a muscle biopsy (quadriceps) before and after the intervention in order to explore protein and mRNA levels of the mTOR pathway, which may be involved in sarcopenia.

DETAILED DESCRIPTION:
Age-related sarcopenia is a common situation defined by muscle mass and function loss in an otherwise healthy elderly person. Epidemiological data from the USA show 49% of men and 72% of women to suffer from sarcopenia. Few data is available on the French population. Sarcopenia is associated with increased morbidity, mortality, disability and reduced resistance to metabolic stress. Resistance training and nutrition are two non-pharmaceutical methods that may be able to prevent several age-related condition.

The aim of this study is to assess the effects of resistance training, associated or not with oral nutritional supplements, on skeletal muscle mass (expressed as skeletal muscle mass index) in sarcopenic subjects. This is a prospective randomised controlled single-centre study that will last two years, three months for a participant.

200 healthy elderly (70-80 years old) subjects will be screened for sarcopenia by dual energy X-ray absorptiometry. 128 sarcopenic subjects will be randomized into 4 groups:

* group 1: controls
* group 2: oral nutritional supplement (260 kcal and 20 g protein per day)
* group 3: resistance training (3 times per week)
* group 4: oral nutritional supplement + resistance training

Every subject will be assessed at the beginning and at the end of 12 weeks of intervention on:

* muscle mass (DXA)
* muscle function (dynamometers)
* hormonal (testosterone, GH, IGF-1, cortisol) and inflammatory (IL-6, TNF-alpha) profiles
* food intake. Ten subjects in group 4 will undergo a muscle biopsy (quadriceps) before and after the intervention in order to explore protein and mRNA levels of the mTOR pathway, which may be involved in sarcopenia.

We expect to show that sarcopenia can be improved by 12 weeks of resistance training and that this improvement can be potentialized by oral nutritional supplements (with a stimulation of the mTOR pathway), and that oral nutritional supplements alone will affect neither muscle mass nor function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 70 and 80 years
* Stable weight (± 1 kg) during the last three months
* Informed consent signed
* Affiliated with the French Sécurité Sociale Non-inclusion criteria
* Chronic cachectic condition: cancer, chronic respiratory failure, advanced organ failure, hyperthyroidism, rheumatoid arthritis, AIDS, type 1 diabetes
* Drugs affecting muscle mass (e.g. steroids)
* Condition (clinical or EKG) significantly affecting physical capacities and/or contra-indicating resistance training
* Habitual practice of resistance training
* Habitual intake of nutritional supplements
* Known coagulation disorders (for muscle biopsy)
* Known allergy to lidocaine (for muscle biopsy)

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
muscle mass (DXA) | D0 and after 12 weeks

SECONDARY OUTCOMES:
muscle function (dynamometers), hormonal (testosterone, GH, IGF-1, cortisol) and inflammatory (IL-6, TNF-alpha) profiles, food intake, ± muscle biopsy. | D0 and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Schneider, PU PH, Principal Investigator — Department of Gastroenterology
Locations (1):
- Department of gastroenterology, Department of Gerontology, Nice, France